CLINICAL TRIAL: NCT06381310
Title: Ultrasound-guided Cannulation of Difficult Hemodialysis Arteriovenous Access: A Randomized Controlled Trial
Brief Title: Ultrasound-guided Cannulation of Difficult Hemodialysis Arteriovenous Access
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Bei-Hu Branch (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202310077DINB
Record Dates: First submitted 2024-04-09; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-02

CONDITIONS: Successful Cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided group (Experimental)
  Interventions: Device: asus-handheld-ultrasound LU710L
- control group (No Intervention)

INTERVENTIONS:
Device: asus-handheld-ultrasound LU710L — Ultrasound-guided group:The nurse uses ultrasound-guide injection. control group: After physical assessment by the nurse, the injection will be carried out according to the conventional injection plan.
  Arms: Ultrasound-guided group

SUMMARY:
Patients with ESRD are able to maintain life by undergoing renal replacement therapy, including hemodialysis (HD), peritoneal dialysis (PD) or kidney transplantation. HD continues to be the primary option. Arteriovenous fistula (AVF) and arteriovenous graft (AVG) are the common access sites for hemodialysis (HD) patients. AVF is the best access for dialysis , which is known as the lifeline of hemodialysis patients, but requires 6 to 8 weeks to maturate. Long-term use of an AVF for dialysis requires the ability of the dialysis staff to cannulate it successfully with large-bore needles thrice weekly. With increasing AVF prevalence as well as aging and more obese populations in the developed world, increasing numbers of difficult-to-cannulate AVFs are being encountered in practice.

Traditionally, after maturation, cannulation of new AVF/AVG was performed by trained renal nurses through physical examination, namely listening to bruits and feeling for thrills to guide needle placement, known as "blind" cannulatio. However, physical examination is not reliable for first and difficult access cannulation (e.g., small or partial stenosis, deep-seated AVF/AVG, presence of clots, after multiple failed attempts with hematoma /swelling, and/or immature access with small vessel caliber), rendered higher rate of cannulation failure and lower AVF and AVG survival. Unfortunately, cannulation failure result in access damage, vessel intimal lining damage leading to stenosis, thrombosis, or aneurysm formation contributing to AVF failure, treatment delay and increased requirement for central venous access devices (CVAD). Patients with early AVF failure have much higher mortality risk, particularly if they are older and female. Van Loon et al. revealed that up to 90% of the first cannulation had complications (i.e., infiltration including hematoma formation and missed cannulation). With a high rate of AVF maturation failure (38-60%) in general, cannulation failure may be avoidable if a more in-depth assessment was done before the attempt.

Ultrasound (US) guided cannulation effective in identifying access location and patency. Roshan et al. reported a case study on bedside ultrasonography for AVF cannulation. The study showed decreased cannulation failure, vessel wall damage, thrombosis, and hematoma formation risks also reduced missed cannulation and increased staff confidence in performing cannulation.

Therefore, this study aims to explore the effects of ultrasound technology on arteriovenous access successful cannulation for patients with end-stage kidney disease to provide reliable research integration evidence as the basis for future clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Those who can undergo the first arteriovenous canal puncture after being evaluated by a physician more than 8 weeks after surgery.
2. The puncture has failed more than 2 times, and there are bruises or hematomas around the arteriovenous and venous vessels.
3. Arteriovenous and venous ducts Ultrasonic detection of arteriovenous and venous ducts ≧0.4, the depth of blood vessels from the skin is 0.4-0.7 cm.
4. The patient has clear consciousness and normal cognitive and communication abilities.

Exclusion Criteria:

1. Under 20 years old.
2. Complex pathways assessed by physicians as having a high risk of complications (diameter ≤ 0.4 cm or depth of blood vessel from skin ≥ 0.8 cm).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
cannulation success rate | 12 times

SECONDARY OUTCOMES:
cannulation satisfaction | 12 times
  Conduct a survey using a self-designed satisfaction questionnaire.Assess satisfaction using Likert scoring criteria. Rate satisfaction on a scale of 0 to 5, with 5 being the highest and 0 being the lowest.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Bei-Hu Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No